CLINICAL TRIAL: NCT04836429
Title: Utilizing Photodynamic Therapy to Amplify the Response to Immunotherapy in Patients With Non-Small Cell Lung Cancer (NSCLC) With Pleural Disease or Malignant Pleural Mesothelioma (MPM) - Phase I Study
Brief Title: Photodynamic Therapy to Amplify the Response to Immunotherapy in Patients With Non-small Cell Lung Cancer With Pleural Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 767720
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Lung Non-Small Cell Carcinoma; Pleural Disorder
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pleural Diseases | interventions — Dihematoporphyrin Ether; Trioxsalen; Thoracic Surgery, Video-Assisted; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment (porfimer sodium, photodynamic therapy) (Experimental): Patients receive porfimer sodium IV over 3-5 minutes 24-48 hours prior to standard of care VATS, followed by photodynamic therapy
  Interventions: Drug: Porfimer Sodium; Procedure: Video-Assisted Thoracic Surgery; Drug: Photodynamic Therapy; Device: Intraoperative PDT

INTERVENTIONS:
Drug: Porfimer Sodium — Given IV
  Other Names: 87806-31-3; CL-184116; Dihematoporphyrin Ester; Photofrin II
Procedure: Video-Assisted Thoracic Surgery — Undergo VATS
  Other Names: VATS
Drug: Photodynamic Therapy — Undergo photodynamic therapy
  Other Names: PDT
Device: Intraoperative PDT — Subjects will receive one course of light therapy at the time of surgery
  Other Names: intra-operative photo dynamic therapy

SUMMARY:
This phase I trial evaluates the side effects of intraoperative photodynamic therapy with porfimer sodium in enhancing the response to immunotherapy with an immune checkpoint inhibitor drug in patients with non-small cell lung cancer with pleural disease. Photodynamic therapy is a technique that that works by combining a photosensitizing agent (porfimer sodium in this trial) and an intense light source to kill tumor cells. Photodynamic therapy may decrease the patients' symptoms and improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (NSCLC) with pleural disease and PDL1 expression < 50% or histologically confirmed diagnosis of malignant pleural mesothelioma not candidates for macroscopic complete resection
* Adequate blood tests 14 days prior to intraoperative PDT and with values within the ranges specified below.

  * Hemoglobin ≥ 9.0 g/L
  * Absolute neutrophil count ≥ 1.5 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (except participants with Gilbert's Syndrome, who are eligible with bilirubin ≤ 2.5 ULN)
  * Alanine transaminase ≤ 2.5 xupper limit of normal (ULN), unless liver metastases or invasion are present, in which case it must be ≤ 5 x ULN
  * Aspartate aminotransferase ≤ 2.5 x ULN, unless liver metastases or invasion are present, in which case it must be ≤ 5 x ULN
* The patient is on standard of care immunotherapy or combination of chemotherapy and immunotherapy with no evidence of progression or a candidate for chemoimmunotherapy as determined by the treating medical oncologist. Eligible patients that are currently on standard of care treatment will have the systemic therapy paused for 4-6 weeks prior to the surgery and intraoperative PDT and will resumed within 4-12 weeks after surgery following standard of care timeframe utilized for restarting systemic therapy after major surgical procedures to ensure adequate post-op recovery and tissue healing.
* Age >= 18 years old
* Life expectancy of at least 12 weeks.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) score of 0 - 1
* Subjects of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for 6 months after surgery. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* The subject must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent prior to receiving any study related procedure
* Platelet count < 100,000

Exclusion Criteria:

* Patients who received chemotherapy, chemoimmunotherapy or radiotherapy within <4 weeks (6 weeks for nitrosoureas or mitomycin C) or those who have not recovered from reversible adverse events prior to the scheduled surgery and intraoperative PDT.
* Patients with untreated or symptomatically unstable treated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with treated and stable brain metastases (at least 28 days from last radiotherapy treatment) are eligible as long as steroids are not required for symptom management
* Patients with porphyria, or with known hypersensitivity to porphyrins or porphyrin-like compounds

  * Absolute neutrophil count < 1500
  * Left ventricular ejection fraction (LVEF) < lower level of normal (LLN)
  * Total bilirubin > 2 mg/dL
  * Creatinine clearance < 60 mL/min (Cockcroft Gault equation)
  * Alkaline phosphatase (hepatic) > 3 times the upper normal limit (SGPT) > 3 times the upper normal limit
  * NOTE: Roswell Park clinical lab blood chemistry is performed on plasma unless otherwise indicated
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female subjects
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the subject an unsuitable candidate to receive porfimer sodium such as active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g. colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included
  * Patients with celiac disease controlled by diet alone
* Patients with Hepatitis B, hepatitis C or human immunodeficiency virus (HIV). Exceptions include past or resolved Hepatitis B (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) and patients positive for hepatitis C (HCV) antibody if polymerase chain reaction is negative for HCV RNA. HIV testing is not required in absence of clinical suspicion of HIV
* Received an investigational agent within 30 days prior to enrollment
* History of, or active autoimmune disorder, requiring systemic steroids or immunosuppressive agents. Exceptions allowed: patients with autoimmune dermatologic conditions not requiring systemic steroids or immunosuppressive agents (e.g. vitiligo, eczema, etc.), endocrine-related autoimmune conditions receiving appropriate hormonal supplementation. Use of immunosuppressant drugs such as steroids, azathioprine, tacrolimus, cyclosporine, etc. is not permitted within 4 weeks before recruitment (exception allowed is use of steroids as hormone replacement therapy or as supportive medication e.g. anti-emesis, contrast allergy, pre-medication, etc. or other short-course therapy less than 2 weeks continuously within 4 weeks of study treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-02-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events (SAE) | 28 days post study-related immunotherapy
  Will be determined by recording the occurrence of SAE during the first 28 days post study-related immunotherapy. The SAE will be evaluated using the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | assessed up to 1 year
  Will utilize Kaplan-Meier curves to descriptively examine dose level differences and generate summary statistics.
Overall survival (OS) | assessed up to 1year
  Will utilize Kaplan-Meier curves to descriptively examine dose level differences and generate summary statistics.
Changes in the immune phenotype of peripheral blood CD8+ T cells | Baseline up to 1year
  Will be analyzed using a repeated measures analysis-of-variance (ANOVA) model with a factor for dose level time and a dose level by time interaction.
Changes in platelet-to-lymphocyte ratio | Baseline up to 1 year
  Will be analyzed using a repeated measures ANOVA model with a factor for dose level, time and a dose level by time interaction.

CONTACTS AND LOCATIONS:
Overall Officials: • Saikrishna Yendamuri, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No